CLINICAL TRIAL: NCT04096807
Title: Perioperative and Non-invasive Estimation of Mean Left Atrial Pressure From Transesophageal Echocardiography Measures of Pulmonary Vein Diameter and Collapsibility in Cardiac Surgery: a Prospective Study
Brief Title: Pulmonary Vein Diameter and Collapsibility Measured by TEE to Predict Elevated Left Atrial Pressure in Cardiac Surgery
Acronym: POGETO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0258
Record Dates: First submitted 2019-08-08; First posted 2019-09-20 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Elevated Left Atrial Pressure
Keywords: Pulmonary wedge pressure; Atrial pressure; Left ventricle; Left ventricular function; Left atrial function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard TEE exam including measurement of left upper pulmonary vein diameter and collapsibility, compared with PCWP measured continuously by a pulmonary arterial catheter — TEE takes part of the standard perioperative hemodynamic monitoring in cardiac surgery. Patients enrolled in the study are also monitored by a pulmonary arterial catheter

SUMMARY:
Left atrial pressure (LAP) is a crucial hemodynamic parameter during cardiac surgery. Elevated LAP leads to pulmonary edema and other cardiopulmonary complications. The pulmonary capillary wedge pressure (PCWP) measured by a pulmonary arterial catheter (PAC) is the gold-standard method to estimate LAP. However, the placement of a PAC is an invasive procedure associated with adverse events. Transesophagial echocardiophy (TEE) is a non-invasive method to estimate LAP during cardiac surgery. Pulsed Doppler mitral flow, pulmonary vein flow, tricuspid regurgitation peak flow and left atrial volume are validated parameters to estimate LAP. Nevertheless, these parameters are not always valid in cardiac surgery, mainly because of mitral valve pathology or prothesis.

As the diameter and collapsibility of inferior vena cava is the recommended method for non-invasive right atrial pressure assessment in patients under mechanical ventilation, the investigators made the hypothesis that diameter and collapsibility of the pulmonary veins could be an additional method to estimate LAP during cardiac surgery. This has never been investigated in cardiology or cardiac surgery.

In this prospective study, pulmonary vein diameter and collapsibility will be correlated to invasive PCWP to assess LAP perioperatively in 30 patients undergoing cardiac surgery

DETAILED DESCRIPTION:
The evaluation of left ventricle filling pressures (LVFP) perioperatively in cardiac surgery could be challenging. This is particularly relevant after separation from cardiopulmonary bypass because the hemodynamic state is dynamic, with changes in heart rate, loading conditions, and deterioration in diastolic function being common. Elevated LVFP leads to pulmonary edema, arrhythmia, pulmonary hypertension and RV failure.

To estimate the LVFP, the gold standard method is the pulmonary capillary wedge pressure (PCWP) measured by a pulmonary arterial catheter (PAC). However, placement of a PAC is an invasive procedure associated with adverse events.

Recommandations released by the American Society of Echocardiography for the evaluation of left ventricular diastolic function pointed out some difficulties concerning the evaluation of elevated LAP perioperativly in cardiac surgery. The commonly used parameters, such as the mitral pulsed Doppler flow, could be faulted by mitral valve regurgitation, atrial fibrillation, or fast changes in loading conditions. In cardiac surgery, additional diagnostic methods are needed to diagnose elevated LVFP.

In the right heart, measurements of the inferior vena cava diameter and collapsibility index are recommended for the evaluation of the right atrial pressure. Since it has been previously described that alterations of the pulmonary vein Doppler flow are correlated with elevated LAP, pulmonary vein diameter dilatation or lack of collapsibility have never been investigated as a marker of elevated LAP, neither in cardiology nor in cardiac surgery.

In this study, the investigators made the hypothesis that pulmonary vein diameter increase when LAP increase (in the absence of confounding factors, such as pulmonary vein stenosis or mitral regurgitation directed toward the pulmonary vein). In the same way,the investigators hypothized that cyclic variations of pulmonary vein diameter under mechanical ventilation decrease when the LAP increase. The ventilation parameters will be standardized.

The investigators will conduct a prospective study in the Department of cardiothoracic anesthesiology and critical care medicine, at the Montpellier University Hospital. Patients scheduled for an elective cardiac surgery and requiring pulmonary arterial catheter monitoring will be enrolled. The TEE standardized protocol will be performed three times, before and after cardiopulmonary bypass, and one-hour postoperatively in ICU. The mean PCWP, the standard method for measuring the LAP, will be recorded simultaneously by the pulmonary arterial catheter. For patients with atrial fibrillation, measurements will be averaged from 10 consecutive cycles.

The main objective is to correlate left upper pulmonary vein diameter and collapsibility with invasive PCWP. We have chosen to analyze the LUPV as the main marker because the LUPV is the easiest to measure among the four pulmonary veins in our clinical practice. Secondary objectives are to explore the correlation between the recommanded LAP echocardiographic parameters and the PCWP ; and to compare the area under curve (AUC) of all echocardiographic parameters to define which parameter has the best predictive value to diagnose elevated LAP. An elevated LAP is defined by a PCWP greater than 18 mmHg.

The study protocol has been approved by the Institutional Rview Board under the number 2019_IRB-MTP_05-21. The IRB waived the need for the investigator to obtain signed consent forms. We have planned to include 30 patients in this study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 18 years or more,
* Scheduled for an elective cardiac surgery at the Montpellier University Hospital,
* Requiring a pulmonary arterial catheter monitoring due to the complexity of cardiac surgery or severe cardiopulmonary comorbidities.

Exclusion Criteria:

* Failure of the pulmonary artery catheterization,
* Failure of PCWP measurement,
* Failure of TEE measure of the left upper pulmonary vein diameter and collapsibility,
* Refusal to participate expressed secondarily.

Non-inclusion criteria :

* Cardiac transplantation,
* Left ventricule assist device,
* Pulmonary vein stenosis,
* Contraindications to TEE or PAC,
* Refusal to participate,
* Patient under juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to the Montpellier University Hospital for cardiac surgery requiring perioperative TEE and pulmonary arterial catheter monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
left upper pulmonary vein diameter (in millimeters) measured by transesophageal echocardiography, compared to the contemporary measure of left atrial pressure by pulmonary arterial catheter. | Pre-cardiopulmonary bypass (15 min before bypass)
  The left upper pulmonary vein (LUPV), which enters the left atrium (LA) just lateral to the LA appendix (LAA) from an anterior to posterior trajectory, can be examined in the mid-esophageal (ME) view at 40 - 60° by slightly withdrawing and turning the probe to the left to expose the superior and lateral aspect of the LA (where the LAA is seen). The LUPV is superior (in the display) to the LAA and separated by the Coumadin ridge.
  Maximal and minimal LUPV diameters will be measured (using a 10 cycle video-loop) and the collapsibility index will be calculated as the ratio : (maximum diameter ¬¬- minimum diameter) / (maximum diameter).
  These echocardiographic views are part of the standard TEE exam and performed with Philips® Epiq™ 7 ultrasound machines.
left upper pulmonary vein diameter (in millimeters) measured by transesophageal echocardiography, compared to the contemporary measure of left atrial pressure by pulmonary arterial catheter. | Post-cardiopulmonary bypass (15 min after bypass)
  The left upper pulmonary vein (LUPV), which enters the left atrium (LA) just lateral to the LA appendix (LAA) from an anterior to posterior trajectory, can be examined in the mid-esophageal (ME) view at 40 - 60° by slightly withdrawing and turning the probe to the left to expose the superior and lateral aspect of the LA (where the LAA is seen). The LUPV is superior (in the display) to the LAA and separated by the Coumadin ridge.
  Maximal and minimal LUPV diameters will be measured (using a 10 cycle video-loop) and the collapsibility index will be calculated as the ratio : (maximum diameter ¬¬- minimum diameter) / (maximum diameter).
  These echocardiographic views are part of the standard TEE exam and performed with Philips® Epiq™ 7 ultrasound machines.
left upper pulmonary vein diameter (in millimeters) measured by transesophageal echocardiography, compared to the contemporary measure of left atrial pressure by pulmonary arterial catheter. | One hour postoperatively in ICU
  The left upper pulmonary vein (LUPV), which enters the left atrium (LA) just lateral to the LA appendix (LAA) from an anterior to posterior trajectory, can be examined in the mid-esophageal (ME) view at 40 - 60° by slightly withdrawing and turning the probe to the left to expose the superior and lateral aspect of the LA (where the LAA is seen). The LUPV is superior (in the display) to the LAA and separated by the Coumadin ridge.
  Maximal and minimal LUPV diameters will be measured (using a 10 cycle video-loop) and the collapsibility index will be calculated as the ratio : (maximum diameter ¬¬- minimum diameter) / (maximum diameter).
  These echocardiographic views are part of the standard TEE exam and performed with Philips® Epiq™ 7 ultrasound machines.

SECONDARY OUTCOMES:
Measurement of the other pulmonary vein diameters | Pre-cardiopulmonary bypass (15 min before bypass)
  Measurement of the other pulmonary vein diameters (in millimeter) : left lower, right upper, right lower pulmonary veins.
Measurement of the other pulmonary vein diameters | Post-cardiopulmonary bypass (15 min after bypass)
  Measurement of the other pulmonary vein diameters (in millimeter) : left lower, right upper, right lower pulmonary veins.
Measurement of the other pulmonary vein diameters | One hour postoperatively in ICU
  Measurement of the other pulmonary vein diameters (in millimeter) : left lower, right upper, right lower pulmonary veins.
Calculation of collapsibility indexes of left upper and right upper pulmonary veins | Pre-cardiopulmonary bypass (15 min before bypass)
  Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
  - Mitral annulus velocities by Tissue Doppler Imaging. Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
Calculation of collapsibility indexes of left upper and right upper pulmonary veins | Post-cardiopulmonary bypass (15 min after bypass)
  Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
  - Mitral annulus velocities by Tissue Doppler Imaging. Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
Calculation of collapsibility indexes of left upper and right upper pulmonary veins | One hour postoperatively in ICU
  Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
  - Mitral annulus velocities by Tissue Doppler Imaging. Calculation of collapsibility indexes of left upper and right upper pulmonary veins. NB: collapsibility index = (maximal diameter - minimal diameter) / (maximal diameter)
Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function | Pre-cardiopulmonary bypass (15 min before bypass)
  Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function : LUPV Doppler flow (S wave, D wave, Ar wave, expressed in m/s), Pulsed Doppler mitral flow (E wave, Am wave, expressed in m/s, E/A ratio, difference Ar -Am), Mitral annulus velocities by Tissue Doppler Imaging (e' velocity, a' velocity, exressed in cm/s), Left atrial area (cm2) and left atrial volume (ml), Left atrial 2D-strain (expressed in negative percentage), Tricuspid regurgitation maximal velocity (in m/s), isovolumic relaxation time (in ms)
Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function | Post-cardiopulmonary bypass (15 min after bypass)
  Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function : LUPV Doppler flow (S wave, D wave, Ar wave, expressed in m/s), Pulsed Doppler mitral flow (E wave, Am wave, expressed in m/s, E/A ratio, difference Ar -Am), Mitral annulus velocities by Tissue Doppler Imaging (e' velocity, a' velocity, exressed in cm/s), Left atrial area (cm2) and left atrial volume (ml), Left atrial 2D-strain (expressed in negative percentage), Tricuspid regurgitation maximal velocity (in m/s), isovolumic relaxation time (in ms)
Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function | One hour postoperatively in ICU
  Measurement of the other echocardiographic parameters estimating the LAP or the left ventricle diastolic function : LUPV Doppler flow (S wave, D wave, Ar wave, expressed in m/s), Pulsed Doppler mitral flow (E wave, Am wave, expressed in m/s, E/A ratio, difference Ar -Am), Mitral annulus velocities by Tissue Doppler Imaging (e' velocity, a' velocity, exressed in cm/s), Left atrial area (cm2) and left atrial volume (ml), Left atrial 2D-strain (expressed in negative percentage), Tricuspid regurgitation maximal velocity (in m/s), isovolumic relaxation time (in ms)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Sentenac, M.D, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC